CLINICAL TRIAL: NCT06575868
Title: Continuous Glucose Monitoring in Myo-inositol Supplemented Obese Pregnant Individuals: a Feasibility Pilot Randomized Control Trial
Brief Title: Myo-inositol During Pregnancy to Prevent Gestational Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00005304
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myo-inositol (Experimental)
  Interventions: Dietary Supplement: Myo-inositol
- Placebo myo-inositol (Placebo Comparator)
  Interventions: Dietary Supplement: Myo-inositol placebo

INTERVENTIONS:
Dietary Supplement: Myo-inositol — Patients would begin taking myoinositol upon recruitment
  Arms: Myo-inositol
Dietary Supplement: Myo-inositol placebo — Patients would begin taking placebo upon recruitment
  Arms: Placebo myo-inositol

SUMMARY:
Myoinositol is an insulin-like compound that is present in both plant and animal cells. Humans synthesize it naturally, but it is also obtained in our diet. It works through an intracellular signaling pathway to increase insulin sensitivity. Myoinositol has been used as an over-the-counter (OTC) supplement in the management of polycystic ovarian syndrome due to this effect. Myoinositol has also been shown to improve glycemic profiles in pregnant euglycemic women and well as improve insulin sensitivity in pregnant patients with gestational diabetes mellitus (GDM).

This is a double blind RCT offering myo-inositol or placebo to those who are eligible and enrolled.

ELIGIBILITY:
Inclusion Criteria:

Singleton gestations

Women aged > 18 years and < 45 years

Recruited before 16 weeks gestation

Obese (pre-pregnancy BMI ≥ 30)

Receiving prenatal care at Tufts Medical Center

Planning to give birth at Tufts Medical Center

Can tolerate glucose tolerance test

Willing and able to wear CGM

Willing and able to sign informed consent

Exclusion Criteria:

Multiple gestation

Preexisting diabetes

Taking medications that impact body weight or metabolism (eg metformin)

Inability to tolerate glucose tolerance test

Adults unable to consent (cognitively impaired adults)

Wards of the state

Non-viable neonates

Neonates of uncertain viability

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Eligibility | 1 year
  proportion of screened women who were eligible
Glucose levels | 1 year
  Average glucose levels during CGM monitoring period for those enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller G, Wied S, Crecelius A, Kessler A, Eckel J. Phosphoinositolglycan-peptides from yeast potently induce metabolic insulin actions in isolated rat adipocytes, cardiomyocytes, and diaphragms. Endocrinology. 1997 Aug;138(8):3459-75. doi: 10.1210/endo.138.8.5308. PMID 9231801
- [Background] Croze ML, Soulage CO. Potential role and therapeutic interests of myo-inositol in metabolic diseases. Biochimie. 2013 Oct;95(10):1811-27. doi: 10.1016/j.biochi.2013.05.011. Epub 2013 Jun 10. PMID 23764390
- [Background] Artini PG, Di Berardino OM, Papini F, Genazzani AD, Simi G, Ruggiero M, Cela V. Endocrine and clinical effects of myo-inositol administration in polycystic ovary syndrome. A randomized study. Gynecol Endocrinol. 2013 Apr;29(4):375-9. doi: 10.3109/09513590.2012.743020. Epub 2013 Jan 22. PMID 23336594
- [Background] Scioscia M, Kunjara S, Gumaa K, Gomez Galan AM, McLean P, Rodeck CH, Rademacher TW. Altered urinary release of inositol phosphoglycan A-type in women with gestational diabetes mellitus. Gynecol Obstet Invest. 2007;64(4):217-23. doi: 10.1159/000106494. Epub 2007 Jul 30. PMID 17664885
- [Background] Malvasi A, Casciaro F, Minervini MM, Kosmas I, Mynbaev OA, Pacella E, Monti Condesnitt V, Creanza A, Di Renzo GC, Tinelli A. Myo-inositol, D-chiro-inositol, folic acid and manganese in second trimester of pregnancy: a preliminary investigation. Eur Rev Med Pharmacol Sci. 2014;18(2):270-4. PMID 24488919
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183
- [Background] D'Anna R, Di Benedetto A, Scilipoti A, Santamaria A, Interdonato ML, Petrella E, Neri I, Pintaudi B, Corrado F, Facchinetti F. Myo-inositol Supplementation for Prevention of Gestational Diabetes in Obese Pregnant Women: A Randomized Controlled Trial. Obstet Gynecol. 2015 Aug;126(2):310-315. doi: 10.1097/AOG.0000000000000958. PMID 26241420
- [Background] Fraticelli F, Celentano C, Zecca IA, Di Vieste G, Pintaudi B, Liberati M, Franzago M, Di Nicola M, Vitacolonna E. Effect of inositol stereoisomers at different dosages in gestational diabetes: an open-label, parallel, randomized controlled trial. Acta Diabetol. 2018 Aug;55(8):805-812. doi: 10.1007/s00592-018-1157-4. Epub 2018 May 17. PMID 29774465
- [Background] D'Anna R, Corrado F, Loddo S, Gullo G, Giunta L, Di Benedetto A. Myoinositol plus alpha-lactalbumin supplementation, insulin resistance and birth outcomes in women with gestational diabetes mellitus: a randomized, controlled study. Sci Rep. 2021 Apr 23;11(1):8866. doi: 10.1038/s41598-021-88329-x. PMID 33893377
- [Background] Vitale SG, Corrado F, Caruso S, Di Benedetto A, Giunta L, Cianci A, D'Anna R. Myo-inositol supplementation to prevent gestational diabetes in overweight non-obese women: bioelectrical impedance analysis, metabolic aspects, obstetric and neonatal outcomes - a randomized and open-label, placebo-controlled clinical trial. Int J Food Sci Nutr. 2021 Aug;72(5):670-679. doi: 10.1080/09637486.2020.1852191. Epub 2020 Nov 25. PMID 33238798
- [Background] Farren M, Daly N, McKeating A, Kinsley B, Turner MJ, Daly S. The Prevention of Gestational Diabetes Mellitus With Antenatal Oral Inositol Supplementation: A Randomized Controlled Trial. Diabetes Care. 2017 Jun;40(6):759-763. doi: 10.2337/dc16-2449. Epub 2017 Mar 21. PMID 28325784
- [Background] Kulshrestha V, Balani S, Kachhawa G, Vanamail P, Kumari R, Sharma JB, Bhatla N. Efficacy of myoinositol in treatment of gestational diabetes mellitus in Asian Indian women: A pilot randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2021 May;260:42-47. doi: 10.1016/j.ejogrb.2021.02.017. Epub 2021 Feb 19. PMID 33721623
- [Background] Amaefule CE, Drymoussi Z, Gonzalez Carreras FJ, Pardo Llorente MDC, Lanz D, Dodds J, Sweeney L, Pizzo E, Thomas A, Heighway J, Daru J, Sobhy S, Poston L, Khalil A, Myers J, Harden A, Hitman G, Khan KS, Zamora J, Perez T, Huda MSB, Thangaratinam S. Myo-inositol nutritional supplement for prevention of gestational diabetes (EMmY): a randomised, placebo-controlled, double-blind pilot trial with nested qualitative study. BMJ Open. 2022 Mar 11;12(3):e050110. doi: 10.1136/bmjopen-2021-050110. PMID 35277398
- [Background] Horgan R, Hage Diab Y, Fishel Bartal M, Sibai BM, Saade G. Continuous Glucose Monitoring in Pregnancy. Obstet Gynecol. 2024 Feb 1;143(2):195-203. doi: 10.1097/AOG.0000000000005374. Epub 2023 Sep 28. PMID 37769316
- [Background] Garcia-Moreno RM, Benitez-Valderrama P, Barquiel B, Gonzalez Perez-de-Villar N, Hillman N, Lora Pablos D, Herranz L. Efficacy of continuous glucose monitoring on maternal and neonatal outcomes in gestational diabetes mellitus: a systematic review and meta-analysis of randomized clinical trials. Diabet Med. 2022 Jan;39(1):e14703. doi: 10.1111/dme.14703. Epub 2021 Oct 13. PMID 34564868
- [Background] Santamaria A, Di Benedetto A, Petrella E, Pintaudi B, Corrado F, D'Anna R, Neri I, Facchinetti F. Myo-inositol may prevent gestational diabetes onset in overweight women: a randomized, controlled trial. J Matern Fetal Neonatal Med. 2016 Oct;29(19):3234-7. doi: 10.3109/14767058.2015.1121478. Epub 2015 Dec 23. PMID 26698911
- [Background] Pintaudi B, Di Vieste G, Corrado F, Lucisano G, Giunta L, D'Anna R, Di Benedetto A. Effects of myo-inositol on glucose variability in women with gestational diabetes. Eur Rev Med Pharmacol Sci. 2018 Oct;22(19):6567-6572. doi: 10.26355/eurrev_201810_16073. PMID 30338829
- [Background] D'Anna R, Scilipoti A, Giordano D, Caruso C, Cannata ML, Interdonato ML, Corrado F, Di Benedetto A. myo-Inositol supplementation and onset of gestational diabetes mellitus in pregnant women with a family history of type 2 diabetes: a prospective, randomized, placebo-controlled study. Diabetes Care. 2013 Apr;36(4):854-7. doi: 10.2337/dc12-1371. Epub 2013 Jan 22. PMID 23340885
- [Background] Parker ED, Lin J, Mahoney T, Ume N, Yang G, Gabbay RA, ElSayed NA, Bannuru RR. Economic Costs of Diabetes in the U.S. in 2022. Diabetes Care. 2024 Jan 1;47(1):26-43. doi: 10.2337/dci23-0085. PMID 37909353
- [Background] Baptiste-Roberts K, Nicholson WK, Wang NY, Brancati FL. Gestational diabetes and subsequent growth patterns of offspring: the National Collaborative Perinatal Project. Matern Child Health J. 2012 Jan;16(1):125-32. doi: 10.1007/s10995-011-0756-2. PMID 21327952
- [Background] Nestler JE, Jakubowicz DJ, Reamer P, Gunn RD, Allan G. Ovulatory and metabolic effects of D-chiro-inositol in the polycystic ovary syndrome. N Engl J Med. 1999 Apr 29;340(17):1314-20. doi: 10.1056/NEJM199904293401703. PMID 10219066
- [Background] D'Anna R, Di Benedetto V, Rizzo P, Raffone E, Interdonato ML, Corrado F, Di Benedetto A. Myo-inositol may prevent gestational diabetes in PCOS women. Gynecol Endocrinol. 2012 Jun;28(6):440-2. doi: 10.3109/09513590.2011.633665. Epub 2011 Nov 28. PMID 22122627
- [Background] Unfer V, Carlomagno G, Dante G, Facchinetti F. Effects of myo-inositol in women with PCOS: a systematic review of randomized controlled trials. Gynecol Endocrinol. 2012 Jul;28(7):509-15. doi: 10.3109/09513590.2011.650660. Epub 2012 Feb 1. PMID 22296306
- [Background] Matarrelli B, Vitacolonna E, D'Angelo M, Pavone G, Mattei PA, Liberati M, Celentano C. Effect of dietary myo-inositol supplementation in pregnancy on the incidence of maternal gestational diabetes mellitus and fetal outcomes: a randomized controlled trial. J Matern Fetal Neonatal Med. 2013 Jul;26(10):967-72. doi: 10.3109/14767058.2013.766691. Epub 2013 Mar 1. PMID 23327487
- [Background] Celentano C, Matarrelli B, Pavone G, Vitacolonna E, Mattei PA, Berghella V, Liberati M. The influence of different inositol stereoisomers supplementation in pregnancy on maternal gestational diabetes mellitus and fetal outcomes in high-risk patients: a randomized controlled trial. J Matern Fetal Neonatal Med. 2020 Mar;33(5):743-751. doi: 10.1080/14767058.2018.1500545. Epub 2018 Dec 17. PMID 30558466
- [Background] Esmaeilzadeh S, Ghadimi R, Mashayekh-Amiri S, Delavar MA, Basirat Z. The effect of myo-inositol supplementation on the prevention of gestational diabetes in overweight pregnant women: a randomized, double-blind, controlled trial. Minerva Obstet Gynecol. 2023 Aug;75(4):357-364. doi: 10.23736/S2724-606X.22.05036-9. Epub 2022 Jun 8. PMID 35686634
- [Background] Castorino K, Polsky S, O'Malley G, Levister C, Nelson K, Farfan C, Brackett S, Puhr S, Levy CJ. Performance of the Dexcom G6 Continuous Glucose Monitoring System in Pregnant Women with Diabetes. Diabetes Technol Ther. 2020 Dec;22(12):943-947. doi: 10.1089/dia.2020.0085. PMID 32324061
- [Background] Motuhifonua SK, Lin L, Alsweiler J, Crawford TJ, Crowther CA. Antenatal dietary supplementation with myo-inositol for preventing gestational diabetes. Cochrane Database Syst Rev. 2023 Feb 15;2(2):CD011507. doi: 10.1002/14651858.CD011507.pub3. PMID 36790138